CLINICAL TRIAL: NCT01246583
Title: A PHASE 2A, MULTI-SITE, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL-GROUP STUDY OF THE PILOT EFFICACY, SAFETY, AND PHARMACOKINETICS OF 2 OINTMENT FORMULATIONS OF CP-690,550 IN SUBJECTS WITH MILD TO MODERATE CHRONIC PLAQUE PSORIASIS
Brief Title: CP-690-550 Ointment For Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3921116
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Results first posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-12

CONDITIONS: Psoriasis
Keywords: Multi Site; Randomized; Placebo Controlled; Double Blind; Parallel Group; chronic plaque psoriasis; topical treatment; skin diseases; papulosquamous
MeSH Terms: conditions — Psoriasis; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment Group A (Experimental)
  Interventions: Drug: CP-690,550 Ointment 1
- Treatment Group B (Placebo Comparator)
  Interventions: Drug: Vehicle 1
- Treatment Group C (Experimental)
  Interventions: Drug: CP-690,550 Ointment 2
- Treatment Group D (Placebo Comparator)
  Interventions: Drug: Vehicle 2

INTERVENTIONS:
Drug: CP-690,550 Ointment 1 — 2% CP-690,550 Ointment 1 twice daily for 4 weeks
  Arms: Treatment Group A
Drug: Vehicle 1 — Vehicle 1 twice daily for 4 weeks
  Arms: Treatment Group B
Drug: CP-690,550 Ointment 2 — 2% CP-690,550 Ointment 2 twice daily for 4 weeks
  Arms: Treatment Group C
Drug: Vehicle 2 — Vehicle 2 twice daily for 4 weeks
  Arms: Treatment Group D

SUMMARY:
The study is being conducted to see whether CP-690,550 ointment has potential as a safe and effective treatment for adult patients with mild to moderate chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate chronic plaque psoriasis (psoriasis vulgaris), with the duration of at least 6 months;
* A target plaque of at least 9 sq. cm.

Exclusion Criteria:

* Demonstrates "rebound" or "flare" of chronic plaque psoriasis;
* Non plaque form of psoriasis;
* Currently have or history of psoriatic arthritis;
* Current drug induced psoriasis;
* Currently on systemic therapy or was on systemic therapy for psoriasis within the previous 6 months;
* Currently on phototherapy for psoriasis or was on phototherapy within the previous 3 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-02-16 (Actual); Primary Completion 2011-11-29 (Actual); Study Completion 2011-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (8):
  - Horizon Research Group, Inc., Mobile, Alabama
  - Dermatology Research Associates, Los Angeles, California
  - Expresscare Medical, Los Angeles, California
  - Park Avenue Dermatology, PA, Orange Park, Florida
  - Skin Specialists, PC, Omaha, Nebraska
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Health Concepts, Rapid City, South Dakota
  - Modern Research Associates, PLLC, Dallas, Texas
- Canada (4):
  - K.Papp Clinical Research Inc., Waterloo, Ontario
  - Innovaderm Research Inc, Montreal, Quebec
  - Siena Medical Research, Montreal, Quebec
  - Centre de Recherche Dermatologique du Quebec metropolitain, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Ports WC, Khan S, Lan S, Lamba M, Bolduc C, Bissonnette R, Papp K. A randomized phase 2a efficacy and safety trial of the topical Janus kinase inhibitor tofacitinib in the treatment of chronic plaque psoriasis. Br J Dermatol. 2013 Jul;169(1):137-45. doi: 10.1111/bjd.12266. PMID 23387374
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921116&StudyName=CP-690-550%20Ointment%20For%20Chronic%20Plaque%20Psoriasis

RESULTS

PARTICIPANT FLOW:
Groups:
- 2% CP-690,550 Ointment 1: CP-690,550 2 percent (%) ointment 1, containing a dermal penetration agent, was applied topically to a 300 square centimeter (cm^2) treatment area twice daily at an application coverage of 3 milligram per cm^2 (mg/cm^2) for 4 weeks.
- Vehicle 1: Placebo ointment (Vehicle 1), matched to 2% CP-690,550 ointment 1, containing a dermal penetration agent, was applied topically to a 300 cm^2 treatment area twice daily at an application coverage of 3 mg/cm^2 for 4 weeks.
- 2% CP-690,550 Ointment 2: CP-690,550 2% ointment 2, without a dermal penetration agent, was applied topically to a 300 cm^2 treatment area twice daily at an application coverage of 3 mg/cm^2 for 4 weeks.
- Vehicle 2: Placebo ointment (Vehicle 2), matched to 2% CP-690,550 ointment 2, without a dermal penetration agent, was applied topically to a 300 cm^2 treatment area twice daily at an application coverage of 3 mg/cm^2 for 4 weeks
Period: Overall Study
Arm/Group | 2% CP-690,550 Ointment 1 | Vehicle 1 | 2% CP-690,550 Ointment 2 | Vehicle 2
Started | 23 | 13 | 25 | 10
Completed | 22 | 13 | 24 | 9
Not Completed | 1 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 2% CP-690,550 Ointment 1: CP-690,550 2% ointment 1, containing a dermal penetration agent, was applied topically to a 300 cm^2 treatment area twice daily at an application coverage of 3 mg/cm^2 for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | 2% CP-690,550 Ointment 1 | Vehicle 1 | 2% CP-690,550 Ointment 2 | Vehicle 2 | Total
Number analyzed (Participants) | 23 | 13 | 25 | 10 | 71
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 years | 7 | 5 | 5 | 4 | 21
  45 to 64 years | 12 | 5 | 13 | 6 | 36
  Greater than or equal to 65 years | 4 | 3 | 7 | 0 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 10 | 4 | 28
  Male | 17 | 5 | 15 | 6 | 43

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Target Plaque Severity Score (TPSS) at Week 4
Description: Target plaque was evaluated individually for signs of induration, scaling and erythema. Each of the 3 signs was rated on 5-point severity scale ranged from 0 to 4: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked. The individual signs severity sub scores were summed to calculate TPSS. The total score varied in increments of 1 and ranged from 1 to 12, with higher scores representing greater severity of psoriasis.
Time Frame: Baseline, Week 4
Population: Full analysis set (FAS) included all participants who were randomized to study and received at least 1 dose of investigational drug (CP-690,550 or vehicle). Here Overall Number of Participants Analyzed signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | 2% CP-690,550 Ointment 1 | Vehicle 1 | 2% CP-690,550 Ointment 2 | Vehicle 2
Number analyzed (Participants) | 22 | 13 | 23 | 9
percent change | -53.97 (29.93) | -41.01 (20.29) | -24.26 (33.43) | -17.24 (25.40)

2. Secondary Outcome: Percent Change From Baseline in Target Plaque Severity Score (TPSS) at Weeks 1, 2 and 3
Description: as for outcome 1
Time Frame: Baseline, Weeks 1, 2, 3
Population: FAS included all participants who were randomized to study and received at least 1 dose of investigational drug (CP-690,550 or vehicle). Here Overall Number of Participants Analyzed= participants who were evaluable for this measure. Number Analyzed=participants evaluable for this measure at specified time points for each treatment group.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | 2% CP-690,550 Ointment 1 | Vehicle 1 | 2% CP-690,550 Ointment 2 | Vehicle 2
Number analyzed (Participants) | 22 | 13 | 24 | 9
percent change
  Change at Week 1: number analyzed (Participants) | 19 | 13 | 23 | 9
  Change at Week 1 | -31.00 (28.54) | -25.59 (18.98) | -12.65 (22.19) | -6.39 (23.06)
  Change at Week 2: number analyzed (Participants) | 21 | 12 | 24 | 7
  Change at Week 2 | -46.32 (29.46) | -28.68 (20.72) | -17.26 (27.50) | -10.32 (26.53)
  Change at Week 3: number analyzed (Participants) | 22 | 13 | 21 | 8
  Change at Week 3 | -49.90 (31.92) | -33.12 (18.92) | -26.32 (32.48) | -27.92 (19.07)

3. Secondary Outcome: Change From Baseline in Target Plaque Severity Score (TPSS) of Erythema, Induration and Scaling at Weeks 1, 2, 3 and 4
Description: Target plaque severity was evaluated individually for signs of induration, scaling and erythema. Each of the 3 signs was rated on 5-point severity scale ranged from 0 to 4: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked.
Time Frame: Baseline, Weeks 1, 2, 3, 4
Population: FAS included all participants who were randomized to study and received at least 1 dose of investigational drug (CP-690,550 or vehicle). Number Analyzed=participants evaluable for this measure at specified time points for each treatment group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 2% CP-690,550 Ointment 1 | Vehicle 1 | 2% CP-690,550 Ointment 2 | Vehicle 2
Number analyzed (Participants) | 23 | 13 | 25 | 10
units on a scale
  Baseline: Erythema | 2.52 (0.59) | 2.62 (0.51) | 2.44 (0.51) | 2.50 (0.53)
  Change at Week 1: Erythema: number analyzed (Participants) | 19 | 13 | 23 | 9
  Change at Week 1: Erythema | -0.53 (0.77) | -0.77 (0.73) | -0.26 (0.62) | -0.11 (0.60)
  Change at Week 2: Erythema: number analyzed (Participants) | 21 | 12 | 24 | 7
  Change at Week 2: Erythema | -0.90 (0.83) | -0.83 (0.58) | -0.42 (0.72) | -0.14 (0.69)
  Change at Week 3: Erythema: number analyzed (Participants) | 22 | 13 | 21 | 8
  Change at Week 3: Erythema | -0.95 (0.90) | -1.00 (0.58) | -0.57 (0.87) | -0.75 (0.71)
  Change at Week 4: Erythema: number analyzed (Participants) | 22 | 13 | 23 | 9
  Change at Week 4: Erythema | -1.14 (0.83) | -1.15 (0.69) | -0.61 (0.89) | -0.44 (0.88)
  Baseline: Induration | 2.52 (0.67) | 2.46 (0.52) | 2.28 (0.46) | 2.40 (0.52)
  Change at Week 1: Induration: number analyzed (Participants) | 19 | 13 | 23 | 9
  Change at Week 1: Induration | -0.68 (0.82) | -0.38 (0.77) | -0.17 (0.58) | 0.00 (0.50)
  Change at Week 2: Induration: number analyzed (Participants) | 21 | 12 | 24 | 7
  Change at Week 2: Induration | -1.05 (0.80) | -0.58 (0.79) | -0.33 (0.70) | -0.14 (0.38)
  Change at Week 3: Induration: number analyzed (Participants) | 22 | 13 | 21 | 8
  Change at Week 3: Induration | -1.18 (0.73) | -0.69 (0.63) | -0.57 (0.81) | -0.38 (0.74)
  Change at Week 4: Induration: number analyzed (Participants) | 22 | 13 | 23 | 9
  Change at Week 4: Induration | -1.27 (0.70) | -0.92 (0.64) | -0.43 (0.90) | -0.22 (0.67)
  Baseline: Scaling | 2.17 (0.65) | 2.23 (0.60) | 2.08 (0.49) | 2.30 (0.82)
  Change at Week 1: Scaling: number analyzed (Participants) | 19 | 13 | 23 | 9
  Change at Week 1: Scaling | -0.95 (0.85) | -0.69 (0.48) | -0.48 (0.95) | -0.33 (0.71)
  Change at Week 2: Scaling: number analyzed (Participants) | 21 | 12 | 24 | 7
  Change at Week 2: Scaling | -1.24 (0.83) | -0.75 (0.75) | -0.38 (0.77) | -0.43 (0.79)
  Change at Week 3: Scaling: number analyzed (Participants) | 22 | 13 | 21 | 8
  Change at Week 3: Scaling | -1.27 (0.88) | -0.85 (0.99) | -0.67 (1.02) | -0.75 (0.71)
  Change at Week 4: Scaling: number analyzed (Participants) | 22 | 13 | 23 | 9
  Change at Week 4: Scaling | -1.32 (0.89) | -1.00 (0.91) | -0.61 (1.03) | -0.56 (0.88)

4. Secondary Outcome: Percentage of Participants With Treatment Area Overall Severity of Psoriasis Response of "Clear" (0) or "Almost Clear" (1)
Description: Treatment area overall severity of psoriasis is global consideration of the erythema, induration and scaling across all psoriatic lesions, rated separately over the treatment area according to a 5-point severity scale ranged from 0 to 4: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked. The severity scores are summed and averaged after which the total average is rounded to the nearest whole number score to determine the treatment area overall severity of psoriasis score and category. Total possible score range: 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe.
Time Frame: Week 1, 2, 3, 4
Population: FAS included all participants who were randomized to study and received at least 1 dose of investigational drug (CP-690,550 or vehicle). Here, Overall Number of Participants Analyzed= participants who were evaluable for this measure. Number Analyzed=participants evaluable for this measure at specified time points for each treatment group.
Measure: Number; unit: percentage of participants
Arm/Group | 2% CP-690,550 Ointment 1 | Vehicle 1 | 2% CP-690,550 Ointment 2 | Vehicle 2
Number analyzed (Participants) | 22 | 13 | 24 | 9
percentage of participants
  Week 1: number analyzed (Participants) | 19 | 13 | 23 | 9
  Week 1 | 42.11 | 23.08 | 21.74 | 11.11
  Week 2: number analyzed (Participants) | 21 | 12 | 24 | 7
  Week 2 | 52.38 | 33.33 | 29.17 | 28.57
  Week 3: number analyzed (Participants) | 22 | 13 | 21 | 8
  Week 3 | 59.09 | 23.08 | 38.10 | 37.50
  Week 4: number analyzed (Participants) | 22 | 13 | 23 | 9
  Week 4 | 63.64 | 61.54 | 39.13 | 22.22

5. Secondary Outcome: Percentage of Participants Achieving Decrease From Baseline of Greater Than or Equal to 2 Points in Treatment Area Overall Severity of Psoriasis Score
Description: Treatment area overall severity of psoriasis is global consideration of the erythema, induration and scaling across all psoriatic lesions, rated separately over the treatment area according to a 5-point severity scale ranged from 0 to 4: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked. The severity scores are summed and averaged after which the total average is rounded to the nearest whole number score to determine the treatment area overall severity of psoriasis score and category. Total possible score: 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe.
Time Frame: Week 1, 2, 3, 4
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | 2% CP-690,550 Ointment 1 | Vehicle 1 | 2% CP-690,550 Ointment 2 | Vehicle 2
Number analyzed (Participants) | 22 | 13 | 24 | 9
percentage of participants
  Week 1: number analyzed (Participants) | 19 | 13 | 23 | 9
  Week 1 | 15.79 | 0.00 | 0.00 | 0.00
  Week 2: number analyzed (Participants) | 21 | 12 | 24 | 7
  Week 2 | 28.57 | 8.33 | 0.00 | 0.00
  Week 3: number analyzed (Participants) | 22 | 13 | 21 | 8
  Week 3 | 31.82 | 15.38 | 9.52 | 0.00
  Week 4: number analyzed (Participants) | 22 | 13 | 23 | 9
  Week 4 | 36.36 | 23.08 | 17.39 | 0.00

6. Secondary Outcome: Percent Change From Baseline in Target Plaque Area at Week 1, 2, 3 and 4
Description: A tracing of the target plaque on transparent film was used to quantify the target plaque area. The target plaque area was calculated by image analysis (planimetry). At baseline, target plaque area was determined prior to randomization to confirm the target plaque size of at least 9 cm^2.
Time Frame: Baseline, Week 1, 2, 3, 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | 2% CP-690,550 Ointment 1 | Vehicle 1 | 2% CP-690,550 Ointment 2 | Vehicle 2
Number analyzed (Participants) | 20 | 12 | 21 | 8
percent change
  Change at Week 1: number analyzed (Participants) | 14 | 12 | 19 | 8
  Change at Week 1 | -14.26 (34.86) | -11.26 (28.55) | -3.72 (19.18) | -3.50 (7.32)
  Change at Week 2: number analyzed (Participants) | 19 | 11 | 20 | 6
  Change at Week 2 | -22.67 (40.18) | -8.35 (37.19) | -5.52 (22.82) | -18.72 (22.18)
  Change at Week 3: number analyzed (Participants) | 18 | 12 | 18 | 7
  Change at Week 3 | -36.21 (42.22) | -13.52 (42.92) | -4.90 (30.23) | -13.59 (38.56)
  Change at Week 4 | -38.39 (43.76) | -19.61 (49.93) | -8.71 (31.23) | -4.98 (27.05)

7. Secondary Outcome: Itch Severity Item (ISI)
Description: The severity of itch was assessed using a single-item Patient Reported Outcome (PRO). Participants were asked to assess their worst itching due to psoriasis at the treatment area over the past 24 hours on a numeric rating scale ranging from of 0-10 where, 0=no itching and 10=worst possible itching.
Time Frame: Baseline, Week 1, 2, 3, 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 2% CP-690,550 Ointment 1 | Vehicle 1 | 2% CP-690,550 Ointment 2 | Vehicle 2
Number analyzed (Participants) | 23 | 13 | 25 | 10
units on a scale
  Baseline | 4.09 (2.52) | 5.54 (3.10) | 4.36 (2.53) | 6.20 (2.62)
  Week 1: number analyzed (Participants) | 19 | 13 | 23 | 9
  Week 1 | 2.63 (2.54) | 4.69 (3.45) | 3.52 (2.74) | 4.22 (3.31)
  Week 2: number analyzed (Participants) | 21 | 12 | 24 | 7
  Week 2 | 2.24 (2.23) | 3.92 (3.12) | 3.42 (2.57) | 4.71 (3.15)
  Week 3: number analyzed (Participants) | 22 | 13 | 21 | 8
  Week 3 | 2.32 (2.42) | 3.69 (3.30) | 2.86 (2.59) | 3.50 (3.02)
  Week 4: number analyzed (Participants) | 22 | 13 | 23 | 9
  Week 4 | 1.55 (2.04) | 3.38 (2.90) | 2.30 (2.20) | 4.44 (2.88)

8. Secondary Outcome: Change From Baseline in the Treatment Area Itch Severity Item (ISI) at Week 1, 2, 3 and 4
Description: The severity of itch was assessed using a single-item PRO. Participants were asked to assess their worst itching due to psoriasis at the treatment area over the past 24 hours on a numeric rating scale ranging from of 0-10 where, 0=no itching and 10=worst possible itching.
Time Frame: Baseline, Week 1, 2, 3, 4
Population: FAS included all participants who were randomized to study and received at least 1 dose of investigational drug (CP-690,550 or vehicle). Here, Overall Number of Participants Analyzed=participants who were evaluable for this measure. Number Analyzed=participants evaluable for this measure at specified time points for each treatment group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 2% CP-690,550 Ointment 1 | Vehicle 1 | 2% CP-690,550 Ointment 2 | Vehicle 2
Number analyzed (Participants) | 22 | 13 | 24 | 9
units on a scale
  Change at Week 1: number analyzed (Participants) | 19 | 13 | 23 | 9
  Change at Week 1 | -1.47 (2.04) | -0.85 (1.63) | -0.74 (2.22) | -2.00 (3.74)
  Change at Week 2: number analyzed (Participants) | 21 | 12 | 24 | 7
  Change at Week 2 | -1.90 (2.14) | -1.83 (3.24) | -1.00 (2.38) | -1.43 (3.87)
  Change at Week 3: number analyzed (Participants) | 22 | 13 | 21 | 8
  Change at Week 3 | -1.86 (1.91) | -1.85 (2.79) | -1.62 (2.65) | -2.75 (4.17)
  Change at Week 4: number analyzed (Participants) | 22 | 13 | 23 | 9
  Change at Week 4 | -2.64 (1.97) | -2.15 (2.85) | -2.13 (2.65) | -1.78 (3.87)

9. Secondary Outcome: Percentage of Participants in Each Patient Satisfaction With Study Medication (PSSM) Response Category
Description: The PSSM evaluates overall participants satisfaction with the study treatment. Participants response evaluation was based on single 7-point item: 1=very satisfied, 2=somewhat satisfied, 3=slightly satisfied, 4=neither satisfied nor dissatisfied, 5=slightly dissatisfied, 6=somewhat dissatisfied, and 7=very dissatisfied.
Time Frame: Week 4
Population: FAS included all participants who were randomized to study and received at least 1 dose of investigational drug (CP-690,550 or vehicle). Here, Overall Number of Participants Analyzed signifies number of participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | 2% CP-690,550 Ointment 1 | Vehicle 1 | 2% CP-690,550 Ointment 2 | Vehicle 2
Number analyzed (Participants) | 22 | 13 | 25 | 9
percentage of participants
  Very Satisfied | 50.0 | 23.1 | 32.0 | 0.0
  Somewhat Satisfied | 18.2 | 38.5 | 20.0 | 11.1
  Slightly Satisfied | 4.5 | 0 | 12.0 | 11.1
  Neither Satisfied nor Dissatisfied | 13.6 | 15.4 | 4.0 | 11.1
  Slightly Dissatisfied | 0 | 0 | 4.0 | 0
  Somewhat Dissatisfied | 4.5 | 7.7 | 12.0 | 22.2
  Very Dissatisfied | 9.1 | 15.4 | 16.0 | 44.4

10. Secondary Outcome: Number of Participants With Administration Site Adverse Events
Description: An adverse event was any untoward medical occurrence attributed to study drug in a participant who received study drug. Application site adverse event included documentation of any clinically significant local reaction, e.g erosion, vesicles or scabbing.
Time Frame: Baseline up to follow up visit (Day 36-39 after last dose of study treatment) (up to maximum of 9.5 weeks)
Population: Safety analysis set included all participants who received at least one dose of the investigational drug (CP-690,550 or vehicle).
Measure: Count of Participants; unit: Participants
Arm/Group | 2% CP-690,550 Ointment 1 | Vehicle 1 | 2% CP-690,550 Ointment 2 | Vehicle 2
Number analyzed (Participants) | 23 | 13 | 25 | 10
Participants | 1 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Burning/Stinging of Psoriatic or Perilesional Skin in The Treatment Area
Description: Burning/stinging symptoms at the treatment area including target plaque, additional plaque/s within the treatment area (if any) and treated perilesional skin (if any) were queried from the participants and scored by the investigator using a 4-point scale: 0=none; 1=Mild; 2=Moderate; 3=Severe. Except at baseline pre-dosing, burning/stinging was assessed for 2 time periods based on the maximum burning or stinging that the participant has experienced: Immediate (within 5 minutes after application); Persistent (beyond 5 minutes after application).
Time Frame: Baseline, Week 1, 2, 3, 4
Population: FAS included all participants who were randomized to study and received at least 1 dose of investigational drug (CP-690,550 or vehicle).
Measure: Count of Participants; unit: Participants
Arm/Group | 2% CP-690,550 Ointment 1 | Vehicle 1 | 2% CP-690,550 Ointment 2 | Vehicle 2
Number analyzed (Participants) | 23 | 13 | 25 | 10
Participants
  Baseline: None, Immediate Stinging/Burning | 0 | 0 | 0 | 0
  Baseline: Mild, Immediate Stinging/Burning | 1 | 0 | 2 | 1
  Baseline: Moderate, Immediate Stinging/Burning | 0 | 0 | 0 | 0
  Baseline: Severe, Immediate Stinging/Burning | 0 | 0 | 0 | 0
  Baseline: None, Persistent Stinging/Burning | 0 | 0 | 1 | 0
  Baseline: Mild, Persistent Stinging/Burning | 1 | 0 | 1 | 1
  Baseline: Moderate, Persistent Stinging/Burning | 0 | 0 | 0 | 0
  Baseline: Severe, Persistent Stinging/Burning | 0 | 0 | 0 | 0
  Week 1: None, Immediate Stinging/Burning | 0 | 0 | 0 | 1
  Week 1: Mild, Immediate Stinging/Burning | 1 | 2 | 0 | 0
  Week 1: Moderate, Immediate Stinging/Burning | 0 | 1 | 0 | 0
  Week 1: Severe, Immediate Stinging/Burning | 0 | 0 | 0 | 0
  Week 2: None, Immediate Stinging/Burning | 0 | 0 | 0 | 0
  Week 2: Mild, Immediate Stinging/Burning | 1 | 0 | 1 | 2
  Week 2: Moderate, Immediate Stinging/Burning | 0 | 0 | 0 | 1
  Week 2: Severe, Immediate Stinging/Burning | 0 | 0 | 0 | 0
  Week 3: None, Immediate Stinging/Burning | 0 | 0 | 0 | 0
  Week 3: Mild, Immediate Stinging/Burning | 1 | 0 | 1 | 0
  Week 3: Moderate, Immediate Stinging/Burning | 0 | 0 | 0 | 0
  Week 3: Severe, Immediate Stinging/Burning | 0 | 0 | 0 | 0
  Week 4: None, Immediate Stinging/Burning | 0 | 0 | 0 | 0
  Week 4: Mild, Immediate Stinging/Burning | 1 | 0 | 0 | 0
  Week 4: Moderate, Immediate Stinging/Burning | 0 | 0 | 0 | 0
  Week 4: Severe, Immediate Stinging/Burning | 0 | 0 | 0 | 0
  Week 1: None, Persistent Stinging/Burning | 1 | 2 | 0 | 0
  Week 1: Mild, Persistent Stinging/Burning | 0 | 1 | 0 | 0
  Week 1: Moderate, Persistent Stinging/Burning | 0 | 0 | 0 | 1
  Week 1: Severe, Persistent Stinging/Burning | 0 | 0 | 0 | 0
  Week 2: None, Persistent Stinging/Burning | 1 | 0 | 1 | 2
  Week 2: Mild, Persistent Stinging/Burning | 0 | 0 | 0 | 0
  Week 2: Moderate, Persistent Stinging/Burning | 0 | 0 | 0 | 1
  Week 2: Severe, Persistent Stinging/Burning | 0 | 0 | 0 | 0
  Week 3: None, Persistent Stinging/Burning | 1 | 0 | 1 | 0
  Week 3: Mild, Persistent Stinging/Burning | 0 | 0 | 1 | 0
  Week 3: Moderate, Persistent Stinging/Burning | 0 | 0 | 0 | 0
  Week 3: Severe, Persistent Stinging/Burning | 0 | 0 | 0 | 0
  Week 4: None, Persistent Stinging/Burning | 1 | 0 | 0 | 0
  Week 4: Mild, Persistent Stinging/Burning | 0 | 0 | 0 | 0
  Week 4: Moderate, Persistent Stinging/Burning | 0 | 0 | 0 | 0
  Week 4: Severe, Persistent Stinging/Burning | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Draize Score of Perilesional Skin in The Treatment Area
Description: Draize scoring evaluated perilesional skin within treatment area for erythema and presence/absence of other signs and symptoms. Erythema score ranged from 0 to 4 as: 0(no reaction visible), 1(trace reactions- barely perceptible pinkness), 2(mild reaction- readily visible pinkness), 3(moderate reaction- definite redness), 4 (Strong to severe reaction- very intense redness). Letter grade defined as: J(Burning, stinging, itching), E(Edema), P(Papules), V(Vesicles), B(Bulla reaction), S(Spreading), W(Weeping), I(Induration), XC(Additional comments). Superficial observations defined as: G(Glazing), Y(Peeling), C(Scab), D(Hyperpigmentation), H(Hypopigmentation), F(Fissuring), R(Erosion), U(Ulceration), K(Scaling). Erythema and other signs/symptoms with at least 1 participant with Draize Score of Perilesional Skin in the treatment area were reported in this outcome measure.
Time Frame: Baseline, Week 1, 2, 3, 4
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | 2% CP-690,550 Ointment 1 | Vehicle 1 | 2% CP-690,550 Ointment 2 | Vehicle 2
Number analyzed (Participants) | 23 | 13 | 25 | 10
Participants
  Baseline, Erythema: Moderate Reaction | 0 | 0 | 1 | 0
  Baseline, Letter Grade: Burning, Stinging, Itching | 2 | 2 | 2 | 0
  Baseline,Superficial Observation:Hyperpigmentation | 0 | 0 | 1 | 0
  Baseline,Superficial Observation: Scaling-Flacking | 0 | 0 | 2 | 1
  Baseline, Superficial Observation: Glazing | 0 | 0 | 1 | 0
  Week 1, Erythema: Trace Reaction | 0 | 0 | 1 | 0
  Week 1, Erythema: Moderate Reaction | 0 | 0 | 1 | 0
  Week 1, Letter Grade: Burning, Stinging, Itching | 1 | 0 | 0 | 0
  Week 1, Superficial Observation: Peeling | 1 | 0 | 0 | 0
  Week 1, Superficial Observation: Scaling-Flacking | 0 | 0 | 2 | 0
  Week 2, Erythema: Trace Reaction | 0 | 0 | 2 | 0
  Week 2, Letter Grade: Burning, Stinging, Itching | 0 | 1 | 0 | 0
  Week 2, Superficial Observation: Scaling-Flacking | 0 | 0 | 1 | 0
  Week 3, Erythema: Trace Reaction | 1 | 0 | 0 | 0
  Week 3, Letter Grade: Burning, Stinging, Itching | 0 | 0 | 2 | 0
  Week 4, Superficial Observation: Hyperpigmentation | 1 | 0 | 0 | 0

13. Secondary Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure at Week 1, 2, 3, 4
Description: Blood pressure (BP) was measured in duplicate (approximately 5 minutes apart) using a standard calibrated BP measuring device. BP defined as pressure exerted by circulating blood upon walls of blood vessels. Diastolic BP is minimum pressure in arteries, near beginning of cardiac cycle when ventricles are filled with blood. Systolic BP is peak pressure in arteries, near end of the cardiac cycle when ventricles are contracting. Normal blood pressure is less than 120 millimeters of mercury (mmHg) systolic and less than 80 mmHg diastolic. Change=value at week 1, 2, 3, 4 minus value at baseline.
Time Frame: Baseline, Week 1, 2, 3, 4
Population: FAS included all participants who were randomized to study and received at least 1 dose of investigational drug (CP-690,550 or vehicle). Number Analyzed=number of participants evaluable for this measure at specified time points for each treatment groups.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 2% CP-690,550 Ointment 1 | Vehicle 1 | 2% CP-690,550 Ointment 2 | Vehicle 2
Number analyzed (Participants) | 23 | 13 | 25 | 10
mmHg
  Baseline: Diastolic BP | 77.91 (9.87) | 74.81 (9.67) | 75.52 (8.63) | 76.60 (10.86)
  Change at Week 1: Diastolic BP: number analyzed (Participants) | 19 | 13 | 23 | 9
  Change at Week 1: Diastolic BP | -3.18 (7.24) | -2.04 (7.17) | -2.54 (8.32) | -1.94 (7.28)
  Change at Week 2: Diastolic BP: number analyzed (Participants) | 21 | 12 | 24 | 7
  Change at Week 2: Diastolic BP | -1.86 (7.41) | -2.25 (5.89) | -3.63 (9.50) | 0.29 (5.80)
  Change at Week 3: Diastolic BP: number analyzed (Participants) | 22 | 13 | 21 | 8
  Change at Week 3: Diastolic BP | -2.23 (8.09) | -3.81 (9.04) | -0.26 (8.64) | -2.13 (8.70)
  Change at Week 4: Diastolic BP: number analyzed (Participants) | 22 | 13 | 23 | 9
  Change at Week 4: Diastolic BP | -2.16 (7.97) | -1.31 (6.94) | -2.61 (7.28) | -1.06 (6.58)
  Baseline: Systolic BP | 120.57 (14.83) | 115.42 (12.77) | 125.62 (16.26) | 116.05 (15.85)
  Change at Week 1: Systolic BP: number analyzed (Participants) | 19 | 13 | 23 | 9
  Change at Week 1: Systolic BP | -2.29 (8.48) | 3.58 (8.76) | -2.85 (8.20) | 3.39 (7.33)
  Change at Week 2: Systolic BP: number analyzed (Participants) | 21 | 12 | 24 | 7
  Change at Week 2: Systolic BP | -2.24 (12.99) | 0.33 (7.24) | -3.67 (8.96) | -3.07 (5.99)
  Change at Week 3: Systolic BP: number analyzed (Participants) | 22 | 13 | 21 | 8
  Change at Week 3: Systolic BP | -0.73 (12.14) | 0.65 (9.29) | 0.67 (8.62) | -0.81 (11.24)
  Change at Week 4: Systolic BP: number analyzed (Participants) | 22 | 13 | 23 | 9
  Change at Week 4: Systolic BP | -0.55 (10.42) | 2.96 (9.73) | -5.07 (9.04) | 1.06 (9.33)

14. Secondary Outcome: Change From Baseline in Heart Rate at Week 1, 2, 3, 4
Description: Heart (pulse) rate was measured in duplicate (approximately 5 minutes apart) for a minimum of 30 seconds. Heart rate is the number of heartbeats per unit of time, usually per minute. The heart rate is based on the number of contractions of the ventricles (the lower chambers of the heart). Change=value at week 1, 2, 3, 4 minus value at baseline.
Time Frame: Baseline, Week 1, 2, 3, 4
Population: FAS included all participants who were randomized to study and received at least 1 dose of investigational drug (CP-690,550 or vehicle). Number Analyzed=participants evaluable for this measure at specified time points for each treatment groups.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | 2% CP-690,550 Ointment 1 | Vehicle 1 | 2% CP-690,550 Ointment 2 | Vehicle 2
Number analyzed (Participants) | 23 | 13 | 25 | 10
beats per minute
  Baseline | 67.24 (10.64) | 66.77 (6.24) | 66.12 (6.82) | 73.75 (8.54)
  Change at Week 1: number analyzed (Participants) | 19 | 13 | 23 | 9
  Change at Week 1 | 2.21 (9.29) | 3.12 (9.98) | 2.28 (8.31) | 6.39 (8.66)
  Change at Week 2: number analyzed (Participants) | 21 | 12 | 24 | 7
  Change at Week 2 | 2.95 (10.75) | 2.71 (6.18) | 2.04 (7.91) | 0.36 (4.41)
  Change at Week 3: number analyzed (Participants) | 22 | 13 | 21 | 8
  Change at Week 3 | 0.61 (7.96) | 2.27 (8.76) | 4.45 (12.41) | 2.50 (3.92)
  Change at Week 4: number analyzed (Participants) | 22 | 13 | 23 | 9
  Change at Week 4 | 2.39 (7.73) | 2.85 (10.60) | 0.63 (7.08) | -2.00 (3.50)

15. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Findings at Week 4
Description: A single standard supine 12-lead Electrocardiogram (ECG) was performed after the participant had rested quietly for at least 10 minutes. ECG parameters included RR interval, PR interval, QRS complex, QT interval, QTcB (corrected for heart rate using Bazett's formula) interval, and QTcF (corrected for heart rate using Fridericia's formula) interval.
Time Frame: Baseline, Week 4
Population: Safety analysis set included all participants who received at least one dose of the investigational drug (CP-690,550 or vehicle). Here, Overall Number of Participants Analyzed signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | 2% CP-690,550 Ointment 1 | Vehicle 1 | 2% CP-690,550 Ointment 2 | Vehicle 2
Number analyzed (Participants) | 22 | 13 | 24 | 9
milliseconds (msec)
  Baseline: RR Interval | 984.7 (165.17) | 958.4 (120.78) | 962.3 (111.02) | 887.9 (124.81)
  Change at Week 4: RR Interval | -47.7 (80.50) | -21.5 (114.31) | -23.1 (107.99) | -8.8 (78.53)
  Baseline: PR Interval | 165.3 (19.80) | 163.8 (26.10) | 159.0 (22.27) | 170.4 (20.70)
  Change at Week 4: PR Interval | -3.5 (11.89) | 2.0 (10.41) | 1.7 (16.73) | 4.2 (11.90)
  Baseline: QRS Complex | 92.8 (5.94) | 93.8 (9.78) | 95.3 (8.38) | 93.0 (5.83)
  Change at Week 4: QRS Complex | -1.5 (7.33) | -2.8 (9.11) | -1.3 (7.11) | -0.3 (9.45)
  Baseline: QT Interval | 400.2 (21.45) | 400.1 (26.91) | 411.1 (26.46) | 392.3 (19.02)
  Change at Week 4: QT Interval | -2.7 (11.40) | -1.2 (22.42) | -8.1 (27.36) | 2.9 (16.04)
  Baseline: QTcB Interval | 406.3 (24.59) | 409.8 (18.53) | 420.1 (19.96) | 418.6 (26.88)
  Change at Week 4: QTcB Interval | 7.1 (16.83) | 5.8 (15.03) | -2.9 (19.77) | 5.4 (16.80)
  Baseline: QTcF Interval | 404.0 (17.23) | 406.5 (18.16) | 417.0 (19.39) | 409.6 (20.03)
  Change at Week 4: QTcF Interval | 3.6 (12.88) | 3.0 (12.86) | -4.8 (19.62) | 4.3 (14.34)

16. Secondary Outcome: Change From Baseline in Hemoglobin Level at Week 2, 4
Time Frame: Baseline, Week 2, 4
Population: FAS population included all participants who were randomized to the study and received at least one dose of the randomized investigational drug (CP-690,550 or vehicle). Number Analyzed =participants evaluable for this measure at specified time points for each treatment group.
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | 2% CP-690,550 Ointment 1 | Vehicle 1 | 2% CP-690,550 Ointment 2 | Vehicle 2
Number analyzed (Participants) | 23 | 13 | 25 | 10
grams per deciliter (g/dL)
  Baseline | 14.56 (1.34) | 13.68 (1.41) | 14.21 (1.26) | 13.90 (1.29)
  Change at Week 2: number analyzed (Participants) | 21 | 13 | 25 | 9
  Change at Week 2 | -0.20 (0.59) | 0.12 (0.48) | 0.19 (0.52) | -0.06 (0.35)
  Change at Week 4: number analyzed (Participants) | 21 | 13 | 23 | 8
  Change at Week 4 | -0.01 (0.56) | -0.08 (0.66) | -0.02 (0.49) | -0.09 (0.39)

17. Secondary Outcome: Change From Baseline in Platelet and Neutrophil Count at Week 2, 4
Time Frame: Baseline, Week 2, 4
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: 10^3 per cubic millimeter (10^3/mm^3)
Arm/Group | 2% CP-690,550 Ointment 1 | Vehicle 1 | 2% CP-690,550 Ointment 2 | Vehicle 2
Number analyzed (Participants) | 23 | 13 | 25 | 10
10^3 per cubic millimeter (10^3/mm^3)
  Baseline: Platelet | 227.30 (69.97) | 212.85 (58.76) | 233.68 (50.79) | 214.90 (58.67)
  Change at Week 2: Platelet: number analyzed (Participants) | 21 | 13 | 25 | 9
  Change at Week 2: Platelet | 6.38 (20.88) | 6.85 (28.31) | 0.00 (21.37) | 13.00 (15.68)
  Change at Week 4: Platelet: number analyzed (Participants) | 21 | 13 | 23 | 8
  Change at Week 4: Platelet | 1.05 (13.88) | -2.46 (15.33) | -7.30 (23.07) | 2.50 (12.65)
  Baseline: Neutrophil | 3.87 (1.36) | 3.75 (1.06) | 4.71 (1.04) | 3.79 (1.48)
  Change at Week 2: Neutrophil: number analyzed (Participants) | 21 | 13 | 25 | 9
  Change at Week 2: Neutrophil | 0.00 (0.59) | 0.00 (0.57) | 0.06 (0.88) | 0.23 (0.51)
  Change at Week 4: Neutrophil: number analyzed (Participants) | 21 | 13 | 23 | 8
  Change at Week 4: Neutrophil | -0.01 (0.77) | -0.21 (0.41) | -0.34 (0.94) | 0.01 (0.57)

18. Secondary Outcome: Change From Baseline in Creatinine Level at Week 2, 4
Time Frame: Baseline, Week 2, 4
Population: FAS population included all participants who were randomized to the study and received at least one dose of the randomized investigational drug (CP-690,550 or vehicle). Number Analyzed=participants evaluable for this measure at specified time points for each treatment group.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | 2% CP-690,550 Ointment 1 | Vehicle 1 | 2% CP-690,550 Ointment 2 | Vehicle 2
Number analyzed (Participants) | 23 | 13 | 25 | 10
milligram per deciliter (mg/dL)
  Baseline | 1.00 (0.22) | 0.89 (0.19) | 0.93 (0.14) | 0.89 (0.17)
  Change at Week 2: number analyzed (Participants) | 21 | 13 | 25 | 9
  Change at Week 2 | -0.02 (0.06) | -0.01 (0.06) | 0.03 (0.07) | -0.04 (0.09)
  Change at Week 4: number analyzed (Participants) | 21 | 13 | 23 | 8
  Change at Week 4 | -0.01 (0.06) | -0.01 (0.07) | -0.02 (0.07) | -0.00 (0.05)

19. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) and Creatine Kinase (CK) Level at Week 2, 4
Time Frame: Baseline, Week 2, 4
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: international unit per liter (IU/L)
Arm/Group | 2% CP-690,550 Ointment 1 | Vehicle 1 | 2% CP-690,550 Ointment 2 | Vehicle 2
Number analyzed (Participants) | 23 | 13 | 25 | 10
international unit per liter (IU/L)
  Baseline: AST | 24.57 (12.35) | 22.77 (6.69) | 23.04 (14.04) | 21.10 (5.38)
  Change at Week 2: AST: number analyzed (Participants) | 21 | 13 | 25 | 9
  Change at Week 2: AST | -2.00 (7.46) | -1.23 (3.83) | 1.84 (4.59) | -2.00 (3.57)
  Change at Week 4: AST: number analyzed (Participants) | 21 | 13 | 23 | 8
  Change at Week 4: AST | -2.29 (7.18) | -1.08 (3.09) | 0.70 (5.98) | 0.63 (3.46)
  Baseline: ALT | 32.22 (26.77) | 28.08 (16.01) | 24.28 (17.81) | 27.60 (13.37)
  Change at Week 2: ALT: number analyzed (Participants) | 21 | 13 | 25 | 9
  Change at Week 2: ALT | -4.48 (14.88) | -3.54 (4.77) | 2.12 (4.75) | -0.67 (7.00)
  Change at Week 4: ALT: number analyzed (Participants) | 21 | 13 | 23 | 8
  Change at Week 4: ALT | -5.76 (17.67) | -3.23 (5.45) | 0.61 (5.75) | -0.13 (1.96)
  Baseline: CK | 117.91 (67.38) | 106.62 (73.11) | 100.16 (61.20) | 93.10 (32.29)
  Change at Week 2: CK: number analyzed (Participants) | 21 | 13 | 25 | 9
  Change at Week 2: CK | -1.05 (40.05) | -11.00 (17.88) | 13.00 (47.55) | 8.00 (56.44)
  Change at Week 4: CK: number analyzed (Participants) | 21 | 13 | 23 | 8
  Change at Week 4: CK | 4.14 (49.49) | 19.62 (73.16) | -2.13 (25.91) | -6.88 (22.25)

20. Secondary Outcome: Plasma Concentration of CP-690,550
Description: Summary statistics were calculated by setting concentration values below the lower limit of quantification (lower limit of quantification=0.1 nanogram per milliliter [ng/mL]) to zero. Summary statistics were not presented if number of observations above lower limit of quantification (NALQ) = 0.
Time Frame: 0 (predose), 1, 2 and 4-9 hours postdose on Day 29 or early termination
Population: Pharmacokinetic analysis set included all treated participants who had at least one plasma concentration value above the lower limit of quantification.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 2% CP-690,550 Ointment 1 | 2% CP-690,550 Ointment 2
Number analyzed (Participants) | 20 | 23
ng/mL
  0 hours | 0.1336 (0.1499) | 0.0313 (0.0742)
  1 hour | 0.1522 (0.1839) | 0.0434 (0.1083)
  2 hours | 0.1548 (0.2089) | 0.0570 (0.1459)
  4 hours | 0.1514 (0.2244) | 0.0553 (0.1420)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | 2% CP-690,550 Ointment 1 | Vehicle 1 | 2% CP-690,550 Ointment 2 | Vehicle 2
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/13 | 0/25 | 0/10
Other Adverse Events (participants affected / at risk) | 10/23 | 3/13 | 9/25 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2% CP-690,550 Ointment 1 (N=23) | Vehicle 1 (N=13) | 2% CP-690,550 Ointment 2 (N=25) | Vehicle 2 (N=10)
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Application site erythema (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Eye infection viral (Infections and infestations) | 1 | 0 | 0 | 0
Labyrinthitis (Infections and infestations) | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 2 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Nerve compression (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Penis disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.